CLINICAL TRIAL: NCT05876780
Title: A Multicenter, Open-label, Single-dose, Systemic Gene Transfer Study to Evaluate the Safety, Tolerability, and Efficacy of SRP-9003 on Subjects With Limb Girdle Muscular Dystrophy, Type 2E/R4 (β-Sarcoglycan Deficiency)
Brief Title: A Gene Transfer Single Dose Study to Evaluate the Safety, Tolerability and Efficacy of SRP-9003 in Non-Ambulatory and Ambulatory Participants With Limb Girdle Muscular Dystrophy, Type 2E/R4 (Beta-Sarcoglycan [β-SG] Deficiency)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRP-9003-102
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Limb Girdle Muscular Dystrophy
Keywords: Ambulatory; Non-ambulatory; Gene-Delivery; LGMD2E/R4; β-SG deficiency; LGMD; Performance of Upper Limb (PUL)
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SRP-9003 (Experimental): Participants will receive single IV infusion of SRP-9003 on Day 1.
  Interventions: Genetic: SRP-9003

INTERVENTIONS:
Genetic: SRP-9003 — Single IV infusion of SRP-9003
  Other Names: scAAVrh74.MHCK7.hSGCB

SUMMARY:
The primary purpose of this study is to evaluate the safety of SRP-9003 and to quantify expression of β-SG in the skeletal muscle of participants with limb-girdle muscular dystrophy, type 2E/R4 (LGMD2E/R4). The study will include both ambulatory (Cohort 1) and non-ambulatory (Cohort 2) participants.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1 only: Ambulatory per protocol specified criteria. - Cohort 2 only: Non-ambulatory per protocol specified criteria and 4 to 50 years of age.
* Possesses 1 homozygous or 2 heterozygous pathogenic and/or likely pathogenic β-sarcoglycan gene Deoxyribonucleic acid (DNA) (SGCB) gene mutations based on documented clinical findings.
* Ability to cooperate with muscle testing.

Exclusion Criteria:

* Presence of any other clinically significant illness or medical condition, including cardiac, pulmonary, hepatic, renal, hematologic, immunologic, neuromuscular (other than LGMD2E/R4), or behavioral disease, or infection or malignancy or concomitant illness or requirement for chronic drug treatment that in the opinion of the Investigator creates unnecessary risks for gene transfer or a medical condition or extenuating circumstance that, in the opinion of the Investigator, might compromise the participant's ability to comply with the protocol required testing or procedures or compromise the participant's wellbeing, safety, or clinical interpretability.
* Exposure to gene therapy, investigational medication, or other protocol-specified treatment within the protocol specified time limits.
* Any contraindication to use of corticosteroid.

Note: Other inclusion or exclusion criteria could apply.

Ages: 4 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2028-08-28 (Estimated); Study Completion 2028-08-28 (Estimated)

PRIMARY OUTCOMES:
Number of Treatment-Emergent Adverse Events (AEs) and Treatment-Emergent Serious Adverse Events (SAEs) | Baseline up to Month 60
Change from Baseline in β-SG Protein Expression Quantity Assessed by Immunofluorescence (IF) Fiber Intensity at Day 60 | Baseline, Day 60
Change from Baseline in β-SG Protein Expression Quantity Assessed by IF Percent Protein Fibers (PPF) at Day 60 | Baseline, Day 60
Change from Baseline in β-SG Protein Expression Quantity Assessed by Western Blot at Day 60 | Baseline, Day 60

SECONDARY OUTCOMES:
Change from Baseline in β-SG Protein Expression Quantity Assessed by IF Fiber Intensity at Month 24 | Baseline, Month 24
Change from Baseline in β-SG Protein Expression Quantity Assessed by IF Percent Protein Fibers (PPF) at Month 24 | Baseline, Month 24
Change from Baseline in β-SG Protein Expression Quantity Assessed by Western Blot at Month 24 | Baseline, Month 24
Change from Baseline in North Star Assessment for Dysferlinopathy (NSAD) at Month 60 | Baseline, Month 60
Change From Baseline in Time to Rise From the Floor, Time to Complete 100 and 10 meter Walk/Run, and the Timed Stair Ascend 4 Steps Test | Baseline, Month 60
Change from Baseline in Performance of Upper Limb Version 2.0 (PUL 2.0) Score at Month 60 | Baseline, Month 60
Change from Baseline in Ability Captured Through Interactive Video Evaluation (ACTIVE) - Seated Workspace Volume Task at Month 60 | Baseline, Month 60
Cohort 1 (Ambulatory): Change from Baseline in Stride Velocity (95%) and Stair-climbing Velocity (95%) as Assessed by a Wearable Device at Month 60 | Baseline, Month 60
Cohort 1 (Ambulatory): Change from Baseline in Number of Stairs Climbed per Hour as Assessed by a Wearable Device at Month 60 | Baseline, Month 60
Cohort 1 (Ambulatory): Change from Baseline Distance Walked per Hour as Assessed by a Wearable Device at Month 60 | Baseline, Month 60
Cohort 1 (Ambulatory): Change from Baseline in Stride Length (95%) as Assessed by a Wearable Device at Month 60 | Baseline, Month 60
Change from Baseline in Upper Extremity Activity at Month 60 | Baseline, Month 60
Change from Baseline in Angular Wrist Velocity at Month 60 | Baseline, Month 60
Change from Baseline in Vector Genome Copies Using Droplet Digital Polymerase Chain Reaction (ddPCR) in the Target Muscle Tissue | Baseline, Day 60 and Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (2):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - St. Jude Children's Research Hospital, Memphis, Tennessee